CLINICAL TRIAL: NCT01310907
Title: Identify the Genes Polymorphisms Related to Non-familial Bradyarrhythmia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Jan-Yow Chen M.D., China Medical University Hospital
Other Study IDs: DMR99-IRB-315
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Bradyarrhythmia
MeSH Terms: conditions — Bradycardia

GROUPS / COHORTS (3):
- sinus node dysfunction
- Atrioventricular block
- control

SUMMARY:
Bradyarrhythmia, including sinus node dysfunction and atrioventricular block, is a major cause necessitating pacemaker implantation. In contrast to familial bradyarrhythmia known as by mutations at particular ion channels, limited information is available for the mechanistic study in non-familial bradyarrhythmia.

Possible gene polymorphisms related to non-familial bradyarrhythmia were studied. Comparison of multi-locus analysis and single-locus analysis will be analyzed between the cases and controls. Functional studies will perform to clarify the results of association study.

ELIGIBILITY:
Inclusion Criteria:

* The patients with non-familial bradyarrhythmia

Exclusion Criteria:

* Familial bradyarrhythmia Reversible bradyarrhythmia Bradyarrhythmia after open heart surgery and severe organic heart diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The case group include 200 patients and the control group include 200 patients.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-02

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Yow Chen, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Background] Mangrum JM, DiMarco JP. The evaluation and management of bradycardia. N Engl J Med. 2000 Mar 9;342(10):703-9. doi: 10.1056/NEJM200003093421006. No abstract available. PMID 10706901
- See also: Heart Rhythm Society — http://www.hrsonline.org/